CLINICAL TRIAL: NCT05906160
Title: The Reliability and Validity of the PortionSize™ and MyFitnessPal Apps (Study 3: Assessment in Free-living Conditions).
Brief Title: PortionSize Study 3: Assessment in Free-living Conditions
Status: Active, not recruiting | Type: Observational
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Corby K. Martin, Professor, Director, Ingestive Behavior Laboratory, Pennington Biomedical Research Center
Other Study IDs: PBRC 2019-063
Record Dates: First submitted 2023-05-26; First posted 2023-06-15 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Dietary Habits
MeSH Terms: conditions — Feeding Behavior

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The study relies on urine samples, which contain a small amount of DNA that degrades after about 4 weeks. The study will not obtain or analyze any DNA related data. The urine will be analyzed to quantify energy expenditure and by extension energy intake.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The objective is to test the accuracy of the PortionSize™ app and the MyFitnessPal© app at measuring energy intake in free-living conditions, tested against the gold-standard, doubly labeled water. Participants will use PortionSize™ and MyFitnessPal apps in separate periods to test the accuracy of the respective apps.

DETAILED DESCRIPTION:
We will recruit adults to use the PortionSize app and the MyFitnessPal free-living conditions. In a within subjects and randomized, counterbalanced design, the accuracy of the PortionSize and MyFitnessPal apps at estimating energy intake in free-living conditions will be tested against the gold-standard, doubly labeled water (DLW), over two non-consecutive four-day periods that should include at least one weekend day and encompass the same days of the week during each period. Participants will be trained in our clinic to use the apps prior to their use in free-living conditions. We will integrate customizable notifications and reminders to remotely prompt participants to record data, resolve data collection problems, etc. These notifications and reminders utilize Ecological Momentary Assessment (EMA) methodology to maximize data collection protocol adherence by reminding participants to capture and send food information at relevant times.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-62 years
* Body mass index (BMI) 18.5-50 kg/m2
* Ownership of an iPhone model 9 or later, which the participant is willing to use for the study
* Access to Apple ID, password, and email address and willing to use them during the study
* Willing to use data and any accompanying charges as part of study participation
* Willing to complete all study procedures and adhere to study visit timelines
* Willing to be re-contacted for future research and/or follow-up

Exclusion Criteria:

oHave been 6-month weight unstable (gain/loss >5% last 6 months) and/or active weight loss program

* Any cardiometabolic disorder that significantly affects what or how much people eat
* Active cancer diagnosis or treatment that significantly affects what or how much people eat, excluding some melanomas and other cancers
* PBRC employee, as previous reviewers argued that they are not representative of the community (
* 3rd member of the same household to participate (i.e. the 1st and 2nd members of the household cannot participate simultaneously)
* Women who are currently pregnant or breastfeeding (self-reported)
* Diagnosed with an uncontrolled thyroid disorder (controlled ≥ 3 months of medication)
* Have had or plan to have weight loss surgery (gastric band removal may be allowed at PI discretion)
* Consume >28 alcoholic beverages per week
* Anyone severely immunocompromised
* Serious digestive disorders that significantly affect what or how much people eat Fluid imbalance and/or on diuretic
* Follows a diet mainly consisting of foods that study staff deems unquantifiable for this study (i.e., liquid supplements, gluten-free specialty items) or consumes a high quantity of specialty foods
* Any condition or circumstance that, in the judgement of the PIs, couldimpede study completion

Ages: 18 Years to 62 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18-62, males and females.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2023-06-22 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Energy Intake (kcal) | May 2023 through February 2025
  Test the equivalence between PortionSize (and MyFitnessPal) and the criterion measure, which is energy intake assessed with DLW. These analyses will rely on equivalence testing using the Two One-side T-test (TOST) method, as well as Bland and Altman analyses.

CONTACTS AND LOCATIONS:
Overall Officials: John W Apolzan, Ph.D., Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided